CLINICAL TRIAL: NCT02308267
Title: Impaired Secretory IgA and Mucosal Immunity in Cystic Fibrosis: Contribution to Lung Pathology and Impaired Defence Against Bacterial Infection
Brief Title: Impaired Secretory IgA and Mucosal Immunity in Cystic Fibrosis
Acronym: Forton2015
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Other Study IDs: Forton2015
Record Dates: First submitted 2014-12-02; First posted 2014-12-04 (Estimated); Last update posted 2016-02-25 (Estimated); Status verified 2016-02

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Mucosal immunity
MeSH Terms: conditions — Cystic Fibrosis | interventions — Bronchoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Lung explants from end-stage CF and control patients, which were obtained for a reason independent from the study.
  2. Sputum, nasal (fluid) and serum samples from CF patients and controls patients (COPD patients and healthy subjects) will be collected for S-IgA and microbiological assays. Spontaneous sputum will be collected, while nasal fluid will be sampled through nasal lavage.
  3. Endobronchial biopsies and broncho-alveolar lavage will be sampled in some CF patients who must have a general anaesthesia for a reason independent from the study. If possible, nasal and rectal biopsies will also be performed. Control subjects will be patients without evidence of lung disease and who are undergoing narcosis for an independent reason.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cystic fibrosis: Cystic fibrosis patients More than 18 years old DF508/DF508 mutation colonized or not with Pseudomonas aeruginosa
  Interventions: Other: Lung explants; Other: Sputum, nasal fluid and serum; Procedure: Bronchoscopy
- Controls: Controls patients More than 18 years old Without CF Smokers or nonsmokers
  Interventions: Other: Lung explants; Other: Sputum, nasal fluid and serum; Procedure: Bronchoscopy

INTERVENTIONS:
Other: Lung explants — Lung explants from end-stage CF, which were obtained for a reason independent from the study in the Paris (Prof Burgel) and Leuven (Prof Dupont) centres will be analysed for pIgR and IgA expression as well as for Pseudomonas aeruginosa colonization. Some lung explants from control patients will also be obtained from the Leuven centre.
Other: Sputum, nasal fluid and serum — Sputum, nasal (fluid) and serum samples from CF patients and controls patients will be collected (Leuven, Paris, Torino, Verona and Saint-Luc Brussels) for S-IgA and microbiological assays. Spontaneous sputum will be collected, while nasal fluid will be sampled through nasal lavage. Control subjects will consist of COPD patients and healthy subjects (smokers or not).
Procedure: Bronchoscopy — Endobronchial biopsies (EBB) and broncho-alveolar lavage (BAL) will be sampled at the KULeuven centre (Prof Dupont) in some CF patients (homozygous for the DF508 mutation) and colonized or not with Pseudomonas aeruginosa and who must have a general anaesthesia for a reason independent from the study. In these patients, a bronchial endoscopy will be performed during narcosis to take EBB (n=8) and BAL (2x50mL). If possible, nasal and rectal biopsies will also be performed in some patients. Samples will be assessed for pIgR and IgA expression and for primary broncho-epithelial cultures (carried out at the UCL centre, Pr Pilette). Control subjects will be patients without CF and without evidence of lung disease and who are undergoing narcosis for an independent reason at the KULeuven centre.

SUMMARY:
This project entitled "Impaired secretory IgA and mucosal immunity in cystic fibrosis" is a research program which aims to determine, owing to national (KULeuven) and international (Descartes university Paris, university of Torino) collaborations for expertise and access to human material, whether a defect exists for the production of IgA antibodies in the lung from patients with this serious genetic disease. These antibodies line and protect normally the airways, and are secreted through a specific epithelial receptor called pIgR (polymeric immunoglobulin receptor); its expression and regulation will be studied in lung tissue and in cell cultures of the lung epithelium from these patients. The link between the putative IgA defect and chronic bacterial infection with Pseudomonas aeruginosa, which often complicates the evolution of the disease, will also be evaluated ex vivo and in vivo, in an animal model of lung infection.

DETAILED DESCRIPTION:
Impaired secretory IgA and mucosal immunity in cystic fibrosis:

role of CFTR-related epithelial changes in the regulation of pIgR-mediated IgA transcytosis and contribution to lung pathology and impaired defence against bacterial infections.

PROJECT DESCRIPTION Cystic fibrosis (CF) represents the most common lethal autosomal recessive disorder in the white population, mainly affecting the lungs. Twenty-four years after the identification of the gene responsible for the disease, many questions remain, current treatments are symptomatic and it remains a lethal disease. It affects the Cystic Fibrosis Transmembrane Regulator (CFTR) gene, which encodes a protein expressed on the apical membrane of airway epithelial cells, where it acts as a cAMP-dependent chloride channel and regulator of other channels, including the epithelial Na+ channel (ENaC). Mutations of the CFTR (F508del, 70% of cases) either result in malfunction or complete absence of the CFTR protein at the apical membrane, due to protein misfolding and retention in the endoplasmic reticulum. It results in defects in chloride efflux and hydration of the epithelial lining fluid, resulting in abnormally viscous mucus which may obstruct the airways, the intestinal lumen and glandular ducts (e.g. in the pancreas). CFTR dysfunction also leads to pro-inflammatory activation (e.g. through NFkB) of the epithelium, resulting in CXCL8/IL8 release (Sloane et al, 2005) and impaired production of protective factors such as a-defensins. Airway colonization of the airways and lung infections are a hallmark of this disease, in particular with Pseudomonas aeruginosa (PA) that affects 70% of CF patients and is associated with poor clinical outcomes. However, the mechanisms underlying the persistence of pathogens in CF airways, remain largely unclear.

This project aims to investigate whether the production of secretory IgA (S-IgA) is impaired in the CF lung, through which mechanisms, and whether this defect contributes to the pathogenesis of CF by impairing immunoprotection against respiratory pathogens such as PA. S-IgA is a major line of mucosal defense, through so-called immune exclusion of inhaled / ingested antigens and pathogens (Norderhaug et al, 1999). Following synthesis of polymeric (mainly dimeric) IgA by subepithelial mucosal plasma cells, p-IgA is transported across the epithelium by a transcellular routing mediated by the polymeric immunoglobulin receptor (pIgR). P-IgA binds to the pIgR at the basolateral pole of the epithelium, and is transcytosed up to the apical pole, where a proteolytic cleavage releases the extracellular part of the pIgR, called secretory component (SC) which remains bound to p-IgA to form S-IgA. This transport represents the most important transcellular routing in the body (3g/day). S-IgA is mainly produced upon mucosal stimulation by microbial signals acting through Toll-like receptors on epithelial cells and B cells (MacPherson et al, 2008) while cytokines (IFN-g, IL-4, IL-1 or TNF-a) may upregulate pIgR expression and/or transcytosis (see review Pilette et al, 2001a).

A defect of pIgR expression has been identified in smoke-induced chronic obstructive pulmonary disease (COPD) (Pilette et al, 2001b). Reduced pIgR in COPD could be due to degradation by neutrophil-derived serine proteinases (Pilette et al, 2003), as well as to impaired gene transcription (Gohy & Pilette, submitted manuscript). In contrast to COPD, it remains unclear whether pIgR expression is affected in CF, through which mechanisms, and if so, with which consequences in terms of mucosal defense. Our hypothesis is that pIgR expression is reduced in CF epithelia, as a result of CFTR-related epithelial changes, and leads to impaired IgA-mediated immune exclusion of respiratory pathogens, thereby favoring chronic bacterial colonization and lung infections in CF. The specific objectives of this project are as follows:

1. to evaluate pIgR & IgA expression in bronchial tissue from CF patients, as compared to controls. This will be performed both in lung explants from CF patients with end-stage lung disease (11 from KULeuven and 18 from Paris, already collected; as compared to 7 explants from controls and to lung surgical specimens from non-smokers) and in bronchial biopsies (n=8) and BAL (2x50mL) sampled during pre-transplantation bronchoscopies (prospective sampling, KULeuven). Control subjects will be patients without CF and without evidence of lung disease and who are undergoing narcosis for an independent reason at the KULeuven centre. In addition, a series of sputum (from CF and control patients) will also be analyzed. Control subjects will consist of COPD patients and healthy subjects (smokers or not). Moreover, nasosinusal and rectal biopsies from CF will also be obtained, in order to investigate mucosal CF tissues outside of the lung environment. Readouts will consist of pIgR expression at both gene (RT-qPCR) and protein (immunohistochemistry, western blot) levels, as well as for IgA (immunohistochemistry, RT-qPCR for IgA1 and IgA2). In addition, (S-)IgA and SC will be measured in bronchial lavage fluids and in sputum.

   Globally, we expected if possible to analyse 30 explants, 30 endoscopies and 150 sputum.
2. to evaluate S-IgA antibodies to respiratory bacteria in CF airways: The relevance of S-IgA deficiency in CF will be assessed with regard to microbial colonisation of lower airways. First, correlation between low S-IgA levels (both total IgA and pathogen-specific IgA) and colonisation by pathogens - in particular PA - will be tested in sputum and bronchial lavage fluids from CF patients. In addition, in lung explants a regional/spatial relationship between S-IgA defect and PA staining will also be addressed. Second, PA-specific IgA antibodies will be assayed in bronchial lavage and sputum fluids, and correlated to colonisation data.
3. to evaluate the contribution of S-IgA defect to lung pathology in CFTR KO mice: The potential contribution of S-IgA deficiency to CF lung disease will be assessed in vivo, using CFTR KO mice. As these KO mice do not recapitulate the human CF phenotype, we will take advantage of our pilot observation that repeated LPS exposure - which leads to a COPD-like phenotype (Juanita et al, 2002) - results in pIgR/SC downregulation (see "Results obtained"). We will thus evaluate whether pIgR deficiency induced upon chronic LPS exposure promotes in CFTR KO mice the development of a lung pathology with CF features. Accordingly, double (CFTR, pIgR) KO mice could be generated to directly address the contribution of pIgR deficiency to lung pathology in conjunction to CFTR mutation. In addition, a second model mimicking persistent PA infection (Martin et al, 2011) will be used to address the effects of PA in CFTR and/or pIgR KO mice. Beta-eNaC Tg mice have a baseline lung pathology and could also be obtained and infected by a model of PA infection (microbeads, Pr Burgel). Readouts will include histomorphological and biomolecular analyses (inflammatory and cytokine responses), and lung function tests (FlexiVent).
4. to explore mechanisms of pIgR downregulation in the CF epithelium: As CFBE 41o-cell line (expressing wt or mutant F508del CFTR; Bruscia et al, 2002) do not express significant levels of pIgR (see "Results obtained"), primary human bronchial epithelial cells (HBEC) will be used to assess whether pIgR downregulation is maintained in the CF epithelium cultured in vitro. Primary cultures in air-liquid interface (ALI) of HBEC will be carried out from CF patients, as compared to controls (up-and-running protocol in the PI's lab in COPD; cells from EpithelixR will also be used; as well as nasal cells from CF (de Courcey et al, 2012)). ALI cultures allow evaluating cellular functions in a polarized and reconstituted muco-ciliary airway epithelium, either resting or stimulated by LPS and/or IL-1. If pIgR expression is also decreased in the CF epithelium in vitro, it could relate to either the CFTR gene defect and/or to epigenetic memory of the in vivo imprinting of the epithelium by the inflammatory microenvironment. We will thus distinguish these possibilities by using CFTR inhibitors (CFTR-inh172, PPQ-102; Martin et al, 2013). Another post-transcriptional mechanism of pIgR dysfunction include its wrong addressing to the cell membrane: the relationship between disturbed expression of each receptor (apical CFTR, basal pIgR) will be evaluated. Readouts will include pIgR expression assessed by immunostaining (of filters) and western blot, and by RT-qPCR. The function of the pIgR will be tested by measuring the capacity of the ALI epithelium to transcytose dimeric IgA from the basolateral to the apical compartment. Membrane addressing of CFTR (apical) and pIgR (basal) will be studied by confocal microscopy.

ELIGIBILITY:
Inclusion Criteria:

CF: adult CF patients (from age 18) with a classical clinical phenotype related to DF508/DF508 mutation, and colonized or not with Pseudomonas aeruginosa

Exclusion Criteria:

* <18 years
* other chronic lung diseases except COPD as a specific control subgroup

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: CF patients followed in a CF center (UCL, KUL, Hôpital Cochin, Torino university) Controls patients (healthy volunteers for sputum or patients undergoing lung surgery for another reason).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-11; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of pIgR & IgA expression in bronchial tissue from CF patients, as compared to controls. | 3 years

SECONDARY OUTCOMES:
Evaluation of S-IgA antibodies to respiratory bacteria in CF airways | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Charles Pilette, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (1):
- StLuc, Brussels, Belgium